CLINICAL TRIAL: NCT00335686
Title: Randomised, Prospective Multicentre Clinical Study on the Effect of the Combination of Lopinavir/Rtv + Nevirapine as Maintenance Bitherapy (Without Nucleoside Analogues) in Comparison With a Triple Therapy Including Lopinavir/Rtv + Nucleoside Analogues in HIV-Infected Patients
Brief Title: Study on the Effect of Kaletra + Nevirapine as Maintenance Bitherapy Compared to a Triple Therapy Including Kaletra + Analogues in HIV Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: LLuita Sida Foundation, LLuita Sida Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MULTINEKA
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2007-06

CONDITIONS: HIV Infections
Keywords: Mitochondrial toxicity; Lopinavir-rtv; Nevirapine; DNA mitochondrial/DNA nuclear
MeSH Terms: conditions — HIV Infections | interventions — lopinavir-ritonavir drug combination; Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Lopinavir-rtv (Kaletra): 3 capsules (600 mg)/12 h
  Interventions: Drug: Lopinavir-rtv (Kaletra): 3 capsules (600 mg)/12 h
- 2 (No Intervention): Nevirapine (Viramune): 1 comp (200mg)/12h
  Interventions: Drug: Nevirapine (Viramune): 1 comp (200mg)/12h

INTERVENTIONS:
Drug: Lopinavir-rtv (Kaletra): 3 capsules (600 mg)/12 h — Lopinavir-rtv (Kaletra): 3 capsules (600 mg)/12 h
  Arms: 1
Drug: Nevirapine (Viramune): 1 comp (200mg)/12h — Nevirapine (Viramune): 1 comp (200mg)/12h
  Arms: 2

SUMMARY:
The study aims to evaluate the changes in mitochondrial DNA (mDNA) by means of the mDNA/nuclearDNA (nDNA) ratio as a marker of mitochondrial toxicity following the interruption of nucleoside analogues.

DETAILED DESCRIPTION:
At the moment it is known that mitochondrial toxicity is the main pathogenic mechanism of toxicity associated with nucleoside analogues, including lipoatrophy, which at facial level is a stigmatising factor for patients with HIV infection.

The primary outcome measure of the design of an "NTRI-sparing" bitherapy is to retard the onset of mitochondrial toxicity or reverse it, mainly with regard to the loss of subcutaneous fat or lipoatrophy.

Lopinavir/ritonavir and nevirapine are two antiretrovirals with different mutation patterns and with high antiviral potency. Their combination therefore guarantees antiviral success. The NEKA study endorses efficacy immunologically and virologically (Negredo E. et al, NRTI-sparing regimen. XIV International AIDS Conference. Barcelona 2002. LB PeB9021).

Similarly, the protective effect of nevirapine on lipid metabolism would counteract the negative impact attributed to lopinavir/ritonavir, reducing cardiovascular risk in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years.
2. HIV-1 infected patients.
3. Patients on HAART therapy with PIs or NNRTIs.
4. Patients with an undetectable viral load (<50/80 copies/mL) over the last 6 months (at least 2 determinations separated by 2 months).
5. Hepatic tests < 5 times the normal value.
6. Subject able to follow the treatment period.
7. Women may not be of fertile age (defined as at least one year from menopause or undergoing any surgical sterilisation technique), or must undertake to use a barrier contraceptive method during the study.
8. Signature of the informed consent

Exclusion Criteria:

1. Presence of opportunistic infections and/or recent tumours (< 6 months).
2. Suspicion of resistance or documented resistance to any of the investigational drugs.
3. Suspicion of possible bad adherence.
4. Pregnancy or breastfeeding; refusal to follow reliable contraception over the treatment period.
5. Known allergic hypersensitivity to any of the investigational drugs or any similar drug.
6. Patients participating in another clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2003-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are changes in the mDNA/nDNA ratio at each visit with regard to the baseline visit. | At 24 and 48 weeks with regard to the baseline visit

SECONDARY OUTCOMES:
Study of the efficacy of the therapy with Lopinavir/rtv (3 tablets every 12 h) + Nevirapine (1 tablet every 12 h) in the maintenance of viral suppression and immune recovery in patients on HAART therapy for more than 9 months | At 12, 24, 36 and 48 weeks.
and CV<50 copies/mL over at last 6 months | At 12, 24, 36 and 48 weeks
To determine whether the combination with Lopinavir/rtv +Nevirapine is efficacious in avoiding progression to lipoatrophy/lipodystrophy or else the reversal thereof | At 24 and 48 weeks
To study whether the combination with Lopinavir/rtv +Nevirapine makes it possible to control dyslipidemia associated with the use of Lopinavir/rtv on proving the "lipid-lowering" action of NVP | At 12, 24, 36 and 48 weeks.
To check whether the simplified combination with the standard dose of Lopinavir/rtv with NVP is sufficient to maintain suppression of viral replication. Pharmacokinetic studies (PK) would be performed to estimate this point | At 12, 24, 36 and 48 weeks
To evaluate the tolerance and safety of the combination of Lopinavir-rtv+Nevirapine . | over 48 weeks of treatment
To evaluate treatment adherence and patient quality of life (evaluated by means of the MOS_HIV questionnaire). | At 12, 24, 36 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD,PhD, Principal Investigator — Lluita contra la Sida Foundation-HIV Unit
Locations (24):
- Spain (24):
  - Hospital C. Universitario de Santiago, Santiago, A Coruña
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Can Mises, Ibiza Town, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Sant Pau, Barcelona, Barcelona
  - Hospital de Mataró, Barcelona, Barcelona
  - Hospital de Granollers, Granollers, Barcelona
  - Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital General de Castellón, Castelló, Castellón
  - Hospital de Figueres, Figueres, Girona
  - Hospital de Palamós, Palamós, Girona
  - Hospital C. San Carlos, Madrid, Madrid
  - Hospital Virgen del Toro, Maó, Menorca
  - Hospital Nuestra Señora del Rosell, Cartagena, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital C. Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Central de Asturias, Asturias, Oviedo
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - Hospital Universitario Joan XXIII de Tarragona, Tarragona, Tarragona
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - Hospital Xeral Cies de Vigo, Vigo, Vigo

REFERENCES:
- [Derived] Negredo E, Miro O, Rodriguez-Santiago B, Garrabou G, Estany C, Masabeu A, Force L, Barrufet P, Cucurull J, Domingo P, Alonso-Villaverde C, Bonjoch A, Moren C, Perez-Alvarez N, Clotet B; MULTINEKA Study Group. Improvement of mitochondrial toxicity in patients receiving a nucleoside reverse-transcriptase inhibitor-sparing strategy: results from the Multicenter Study with Nevirapine and Kaletra (MULTINEKA). Clin Infect Dis. 2009 Sep 15;49(6):892-900. doi: 10.1086/605440. PMID 19663689